CLINICAL TRIAL: NCT02507947
Title: SPECTAmel: Screening Patients With Melanoma Tumors for Efficient Clinical Trial Access
Status: Withdrawn | Type: Observational
Why Stopped: Study closed
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-1332
Record Dates: First submitted 2015-07-23; First posted 2015-07-24 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — FFPE block of tumor tissue, blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
SPECTAmel is a standardized, quality-assured molecular screening platform for tumor characterization and storage of human biological material (HBM) for the purpose of integrating new biomarkers into clinical trials and optimizing access of patients to therapeutic biomarker-driven clinical trials. HBM and clinical/pathological data are collected from consenting patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed melanoma of any stage (the steering committee will decide on which stage to include at any particular time point during this trial, this will be communicated appropriately to all participating sites)
* Mandatory availability of adequate human biological material (HBM): FFPE tissue sample from the primary tumor, recurrent tumor, metastasis, obtained at the time of primary surgery/biopsy; minimal amount requested is detailed in the HBM guidelines; if feasible, inclusion of samples taken at any recurrence diagnosed during follow-up is strongly encouraged but optional;
* Age ≥ 18 years;
* At least three months life-expectancy;
* Written informed consent according to ICH/GCP and national/local regulations;
* Absence of any active malignancy, except pT1-2 prostatic cancer Gleason score < 6, or carcinoma in situ of the cervix, in the 5 years before study entry;
* Absence of exclusion criteria like active hepatitis B/C or HIV, second malignancies, no severe organ dysfunction or other comorbidities that may prevent inclusion into clinical trials.
* Central confirmation of human biological material (HBM) adequacy for step 2:
* Centrally performed confirmation of tumor tissue adequacy in terms of quality/ quantity for central screening.

Exclusion Criteria:

* active hepatitis B/C or HIV
* second malignancies
* severe organ dysfunction or other comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathologically confirmed melanoma of any stage
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Primary Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Number of screened patients | 5 years
Number of downstream clinical trials; | 5 years
Number of patients enrolled in the downstream therapeutic trials | 5 years
Number of exploratory/future research projects | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Robert, MD, PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris